CLINICAL TRIAL: NCT04246970
Title: Effects of a Prehabilitation Program in Liver Transplant Candidates Followed by a Posttransplant Training Program
Brief Title: Prehabilitation and Posttransplant Training Program in Liver Transplantation
Acronym: PreLiveR-T
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maria dels Angels Cebria i Iranzo, PT, PhD (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor-Investigator, Maria dels Angels Cebria i Iranzo, PT, PhD, Director research, Hospital Universitario La Fe
Organization: Hospital Universitario La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/0227
Record Dates: First submitted 2020-01-20; First posted 2020-01-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant; Complications; Cirrhosis, Liver; Hepatic Carcinoma
Keywords: Prehabilitation; Therapeutic Exercise; Functional capacity
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular | interventions — Preoperative Exercise; Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Conventional medical care
- Prehabilitation group (Experimental): Conventional medical care and 8 weeks of a Prehabilitation supervised program
  Interventions: Other: Prehabilitation
- Prehabilitation and posttransplant training group (Experimental): Conventional medical care, 8 weeks of a Prehabilitation supervised program and a posttransplant training program.
  Interventions: Other: Prehabilitation; Other: Prehabilitation and posttransplant training program

INTERVENTIONS:
Other: Prehabilitation — Supervised training program of 8-weeks and a frequency of 2 days/week. It includes interval aerobic exercise (5 cycles of 2 minutes at 70 percentage of Watts or heart rate of cardiopulmonary exercise testing (CEPT) and 3 minutes of active rest at 40 percentage; peripheral muscle training and balance exercises in a circuit of 10 phases, 10 to 15 repetitions, from 1 to 3 sets (the participants will work at moderate intensity, no more than 5-6/10 on the modified Borg scale); Inspiratory Muscle Training (IMT) through a threshold loading device [2 sessions / day, 3 sets of 15 repetitions, at 60-70 percentage of the maximum inspiratory pressure (cmH2O)]; ventilatory reeducation by an incentive inspirator based on the vital capacity evaluated in the initial spirometry. Both the aerobic modality and the resistance training, will increase the intensity of work (HR, Watts, Kg or cmH2O) between 2-5 percentage every 2 weeks complying with the principle of training overload.
  Other Names: Interval aerobic exercise, peripheral and respiratory muscle training, balance exercise
  Arms: Prehabilitation and posttransplant training group; Prehabilitation group
Other: Prehabilitation and posttransplant training program — Prehabilitation will be followed by a posttransplant training program. In this, the patient will perform supervised exercise (IIa interval aerobic exercise and resistance training) 2 days / week, and a physical exercise program at home until completing a total of 5 sessions / week in the aerobic modality. In the unsupervised phase (IIb), the patient will continue with the learned physical exercise program, but without supervision, 5 sessions / week (including a minimum of 2 non-consecutive sessions to perform resistance training).
  Other Names: Interval aerobic exercise, peripheral muscle training and balance exercise
  Arms: Prehabilitation and posttransplant training group

SUMMARY:
PreLiveR-T consists of a prospective randomized clinical trial conducted in an adult population that is a candidate for liver transplantation (LT) at the Hospital La Fe Valencia (Spain). The study is structured in three phases: I) Prehabilitation (2 months before LT); II) Training, divided in two successive periods: Supervised training (months 3-6 after LT) and Unsupervised training (6-12 months after LT); III) Long-term follow-up (2 years after LT).

Primary outcomes are related to post-surgery evolution (morbidity and mortality, hospitalization length, etc.). As a secondary outcomes are collected those related to: functional capacity, muscle strength and quality of life.

DETAILED DESCRIPTION:
The main objective is to study the post-surgical impact (post-S) of a Prehabilitation program on candidates for liver transplantation (LT), as well as to study the effects of posttransplant training on the clinical and functional evolution of the recipients. Also this project pretends to assess the influence of functional capacity (FC) improvement on the short and long term post-S evolution of the LT candidates. This is a prospective randomized clinical trial in which three phases follow: Prehabilitation, training and follow-up. The sample will be constituted by 60 candidates for LT, randomized in a control group (CG, n=20), a Prehabilitation group (PG, n=20) and a Prehabilitation-posttransplant training group (PTG, n=20). To conventional care, a Prehabilitation program will be added to the PG and PTG. After the LT, just PTG will follow a posttransplant training program. The long-term follow-up will be extended to 2 years post-LT. The variables under study will be: complications and post-S evolution; FC; quality of life; etc. The individualization of Prehabilitation and posttransplant training program, and also medical control, will ensure safety and offer the potential benefits that these types of programs can provide.

ELIGIBILITY:
Inclusion Criteria:

* Indication of elective liver transplant with favorable cardiorespiratory evaluation that does not contraindicate the transplant.

Exclusion Criteria:

* Any orthopedic, motor, functional, neurological, cognitive or linguistic limitation that prevents the realization of the Prehabilitation program
* Inability to perform psychometric tests
* Esophageal varices not treated with ligature or beta-blockers
* Varicose veins with a high risk of digestive hemorrhage
* Hemoglobin <80 g/l
* Contraindication to weight loading
* Impossibility to comply with the Prehabilitation program (hospital admission, work, geographical location)
* Multi-organ transplantation and liver retransplantation
* Refusal or lacks capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Morbidity | The groups will be assessed from the hospitalization up to 24-months.
  Registry of post-surgical complications according to the Clavien-Dindo classification. Reference: Ann Surg 2004; 240(2):205-13.
Mortality | The groups will be assessed from the hospitalization until the date of death, assessed up to 24-months.
  Registry of mortality
Number of hospitalization days | The groups will be assessed during hospitalization, approximately 7 days.
  Registry of number of days of hospitalization in intensive care unit and ward.
Number of days with supplementary oxygen therapy and/or mechanical ventilation | The groups will be assessed during hospitalization, approximately 7 days.
  Registry of number of days
Progression in the activities of daily life (ADL) | The groups will be assessed during hospitalization, approximately 7 days.
  Days of acquisition, sitting, walking and stairs

SECONDARY OUTCOMES:
Change in functional capacity: measurement of oxygen uptake | The groups will be assessed at four times: at baseline; at week 8; 3-months after LT; and 6-months after LT.
  Cardiopulmonary exercise test following an incremental protocol on ramp with a bicycle ergometer.
Change in functional capacity: 6-minutes walking test (6MWT) | The groups will be assessed at four times: at baseline; at week 8; 3-months after LT; and 6-months after LT.
  6MWT is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6 MWT provides information regarding functional capacity, response to therapy and prognosis. American Thoracic Society (ATS) Statement Guidelines for the Six-Minute Walk Test. Am J Resp Crit Care Med 2002;166(1):111-117
Change in peripheral muscle strength: handgrip strength, quadriceps femoris strength and biceps brachii strength | The groups will be assessed at six times: at baseline; at week 8; 1-month, 3-months, 6-months and 24-months after LT.
  Isometric peripheral muscle strength will be measured using a digital hand dynamometer and the unit of measure is kilograms. References:
  Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall CC, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age and Ageing 2011;40(4):423-9.
  Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996; 76(3):248-59
Change in respiratory strength: maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) | The groups will be assessed at baseline and at week 8.
  Maximum respiratory pressures will be measured using a Respiratory Pressure Meter MicroRPM® and the unit of measure is cmH2O. MIP and MEP are probably the most frequently reported non-invasive estimates of respiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal breathing. Reference: Am J Respir Crit Care Med. 2002;166:531-535
Change in performance on the Short Physical Performance Battery (SPPB) | The groups will be assessed at six times: at baseline; at week 8; 1-month, 3-months, 6-months and 24-months after LT.
  The SPPB is a simple test to measure lower extremity function using tasks that mimic daily activities. The SPPB examines three areas of lower extremity function; static balance, gait speed, and getting in and out of a chair. Static balance is measured in units of time (seconds) and patients are timed holding 3 different stances. Gait speed is measured in time (seconds) to walk 4 meters. Chair sits are measured as the time (seconds) it takes to get up and out of a chair 5 times without using one's arms to assist the exercise. Collectively, the three tests are used to generate a total score (0-12) that reflects a patient's frailty (score of 0) or lack of frailty (score of 12). Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994;49:M85-M94.
Change in muscle mass | The groups will be assessed at six times: at baseline; at week 8; 1-month, 3-months, 6-months and 24-months after LT.
  Bioelectrical impedance analysis will be completed using the Bodystat 1500 MDD, which is a multi-frequency body composition analyzer. Body fat percentage (%) will be compared to lean body mass percentage and total body water percentage to assess sarcopenia and nutritional status.
Change in Quality of life | The groups will be assessed at six times: at baseline; at week 8; 1-month, 3-months, 6-months and 24-months after LT.
  Short-Form Liver Disease Quality of Life (SF-LDQOL) is formed by 9 dimensions: symptoms of the disease, effects of the disease on the activities of daily life, memory/concentration, anxiety, sleep, loneliness, hopelessness, stigma for the disease and sexual functioning. The minimum and maximum values of the scale are 0-100, so that the higher the score, the better health related quality of life (HRQL).

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Cebrià i Iranzo, PT, PhD, Principal Investigator — Hospital Universitari i Politècnic La Fe, Valencia; David Calatayud Mizrahi, MD, PhD, Study Chair — Hospital Universitari i Politècnic La Fe, Valencia; Natalia Cezón Serrano, PT, Study Chair — University of Valencia; Luis Compte Torrero, MD, PhD, Study Chair — Hospital Universitari i Politècnic La Fe, Valencia; Laura Arjona Tinaut, PT, Study Chair — University of Valencia; Rafael López Andújar, MD, PhD, Study Chair — Hospital Universitari i Politècnic La Fe, Valencia; Martín Prieto Castillo, MD, PhD, Study Chair — Hospital Universitari i Politècnic La Fe, Valencia
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Brustia R, Savier E, Scatton O. Physical exercise in cirrhotic patients: Towards prehabilitation on waiting list for liver transplantation. A systematic review and meta-analysis. Clin Res Hepatol Gastroenterol. 2018 Jun;42(3):205-215. doi: 10.1016/j.clinre.2017.09.005. Epub 2017 Nov 20. PMID 29162460
- [Background] Debette-Gratien M, Tabouret T, Antonini MT, Dalmay F, Carrier P, Legros R, Jacques J, Vincent F, Sautereau D, Samuel D, Loustaud-Ratti V. Personalized adapted physical activity before liver transplantation: acceptability and results. Transplantation. 2015 Jan;99(1):145-50. doi: 10.1097/TP.0000000000000245. PMID 25531893
- [Background] Williams FR, Vallance A, Faulkner T, Towey J, Durman S, Kyte D, Elsharkawy AM, Perera T, Holt A, Ferguson J, Lord JM, Armstrong MJ. Home-Based Exercise in Patients Awaiting Liver Transplantation: A Feasibility Study. Liver Transpl. 2019 Jul;25(7):995-1006. doi: 10.1002/lt.25442. Epub 2019 Jun 6. PMID 30859755